CLINICAL TRIAL: NCT03443297
Title: Early Versus Delayed Enteral Feeding for Achieving Full Feeding in Preterm Growth-Restricted Infants: A Randomized Clinical Trial
Brief Title: Early Versus Delayed Feeding in Preterm Growth-Restricted Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Farzana Ahmed, Honorary medical officer, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U1111-1203-7088
Record Dates: First submitted 2018-02-06; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Preterm Infant; IUGR
MeSH Terms: conditions — Premature Birth | interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Feeding group (Experimental): Active ingredient: maternal expressed breast milk Time of initiation of first feeding: 24 to 48 hours of age. Doses: Initially 4 hourly feeding will be started with 0.5 ml and 1 ml expressed breast milk in babies with birth weight <1200 grams and >1200 grams respectively. On the following day 3 hourly, thereafter 2 hourly feeding will be provided in both groups. Gradually amount of feeding will be increased after reaching 2 hourly feeding at the rate of 10 ml/kg/day for initial 10 days then 20ml/kg/day in 2 aliquots till full feeding(150ml/kg/day).For babies with birth weight <1200 gram, rate of feeding advancement 10 ml/kg/day till full feeds. Time of starting first feeding and time to reach full feeding, both will be documented in a questionnaire for each patient.
  Interventions: Other: breast milk
- Late Feeding group (No Intervention): Feeding with maternal breast milk will be given in conventional way

INTERVENTIONS:
Other: breast milk — Feeding with breast milk will be started in early feeding group from 24 to 48 hours of age or in late feeding group, from 48 to 72 hours of age. Initially 4 hourly feeding will be started with 0.5ml and 1 ml expressed breast milk in babies with birth weight <1200 grams and >1200 grams respectively. gradually volume of milk should be increased
  Arms: Early Feeding group

SUMMARY:
The introduction of enteral feeds for preterm, growth restricted infants are often delayed due to concern that early introduction may not be tolerated and may increase the risk of necrotizing enterocolitis. However, prolonged enteral fasting may diminish the functional adaptation of the immature gastrointestinal tract and extend the need for parenteral nutrition with its attendant infectious and metabolic risks. Early introduction of small volumes of milk in the form of Trophic feeding, promote intestinal maturation, may enhance feeding tolerance and decrease the time taken to reach full enteral feeding independently of parenteral nutrition.

A Randomized Trial will be carried out over a period of 12 months in Department of Neonatology of BSMMU. Sample size will be 50(25 in each group). Infants with gestation below 35 weeks, birth weight below the 10th percentile for gestational age, will be randomly allocated by web-based randomization to commence enteral feeds "early," whose feeding will be started from 24 to 48 hours of age or "late," whose feeding will be started from 48 to 72 hours of age. Gradually feeding will be increased. Rate of advancement of feeding will be same for both groups. Primary outcomes will be time to achieve full enteral feeding sustained for 72 hours. Statistical analyses will be performed by using Fisher Exact test and by Student's t test for categorical data and quantitative data respectively. Logistic regression analyses will be performed to determine the role of independent variable.

DETAILED DESCRIPTION:
Eligible infants who will fulfill the inclusion criteria will be divided into two strata "Early feeding group" and " Late feeding group" by computer based randomization after taking informed written consent from parents or responsible caregivers. Feeding will be started in early feeding group from 24 to 48 hours of age or in late feeding group, from 48 to 72 hours of age. Initially 4 hourly feeding will be started with 0.5ml and 1 ml expressed breast milk in babies with birth weight <1200 grams and >1200 grams respectively. On the following day 3 hourly, thereafter 2 hourly feeding will be provided in both groups. Gradually amount of feeding will be increased after reaching 2 hourly feeding at the rate of 10 ml/kg/day for initial 10 days then 20ml/kg/day in 2 aliquots till full feeding(150ml/kg/day).For babies with birth weight <1200 gram, rate of feeding advancement 10 ml/kg/day till full feeds. Any baby who will develop shock (due to sepsis, cardiogenic, hypovolemic etc.) will be excluded and will be replaced by new one in same category as per protocol analysis. Follow up examinations will be done.

ELIGIBILITY:
Inclusion Criteria:

* All growth restricted preterm Infants of both sexes with gestational age 35 weeks or less and birth weight below 10th percentile for gestational age

Exclusion Criteria:

* • Hemodynamically unstable critically ill neonates.

  * Newborn with severe perinatal asphyxia.
  * Newborn with polycythemia requiring exchange transfusion
  * Newborn with major congenital anomalies
  * Syndromic manifestations or chromosomal malformations
  * Suspected inborn errors of metabolism.
  * Any baby who will have proven sepsis with shock or necrotizing enterocolitis will be excluded and will be replaced by new one in same category as per protocol analysis.
  * Any baby who develop shock (due to sepsis, cardiogenic, hypovolemic etc.) will be excluded and will be replaced by new one in same category as per protocol analysis.

Ages: 1 Minute to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of feeding with weight gain pattern | 1 year
  Early achievement of acceptable weight gain 20-25 gram per day

IPD SHARING:
Plan to Share IPD: No